CLINICAL TRIAL: NCT06923488
Title: Phase I/II Study of Leflunomide in Combination With Decitabine for Treatment of Relapsed or Refractory (R/R) Myelodysplastic Syndromes (MDS)
Brief Title: Leflunomide in Combination With Decitabine for Treatment of Relapsed or Refractory Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Konstantinos Sdrimas, Assistant Professor, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2502109808
Record Dates: First submitted 2025-03-25; First posted 2025-04-11 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: relapsed or refractory
MeSH Terms: conditions — Myelodysplastic Syndromes; Recurrence | interventions — Leflunomide; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leflunomide + Decitabine Treatment (Experimental): Participants will receive combination treatment for 12 cycles consisting of 28 days. Utilizing a conventional 3+3 design, Decitabine will be at a dose of 20 mg/m2 and will be administered by intravenous infusion over 1 hour daily for 5 days each 28-day cycle. Leflunomide will have a dose escalation schedule starting at (Level +1) as follows:
  Dose Escalation (Level -2): Leflunomide 10mg once daily by mouth x 14 days/cycle (Level -1): Leflunomide 10mg once daily by mouth x 21 days/cycle (Level +1): Leflunomide 20mg once daily by mouth x 14 days/cycle (Level +2): Leflunomide 20mg once daily by mouth x 21 days/cycle
  Interventions: Drug: Leflunomide 10mg; Drug: Leflunomide 20mg; Drug: Decitabine

INTERVENTIONS:
Drug: Leflunomide 10mg — Leflunomide 10mg tablet
  Other Names: Arava
Drug: Leflunomide 20mg — Leflunomide 20mg tablet
  Other Names: Arava
Drug: Decitabine — Decitabine dose of 20 mg/m2
  Other Names: Dacogen

SUMMARY:
The goal of this interventional clinical trial is to evaluate the safety and tolerability of leflunomide in combination with decitabine as treatment for patients with relapsed or refractory myelodysplastic syndromes (R/R MDS).

The main question this study aims to answer are to evaluate and estimate the maximum tolerated doses and/or biologically active doses of the combination of leflunomide-decitabine in participants.

Decitabine will be administered at a dose of 20 mg/m2 by continuous intravenous infusion over one hour repeated daily for 5 days with repeating cycle every 4 weeks. Leflunomide is administered orally at 10 to 20 mg once daily (without a loading dose) for 14 to 21 days, as part of a 28-day treatment cycle in adult subjects with R/R MDS. After 12 cycles (study duration) responding patients can continue progression with the assigned doses.

DETAILED DESCRIPTION:
This is a phase I/II dose-escalation trial to estimate the activity of leflunomide in combination with decitabine for treatment of relapsed or refractory MDS. Leflunomide will be administered orally daily with decitabine IV for 5 days as part of a 28-day treatment cycle in adult subjects with R/R MDS. Patients who have been previously treated with decitabine will be eligible. The trial will consist of dose escalation to evaluate safety and tolerability of leflunomide in combination with decitabine. There will be no intra-patient dose escalation or reduction. In the event of an RLT, one or both drugs (leflunomide or decitabine) could be withheld at the discretion of the treating physician and on the basis of the expected adverse event. The period for determination of RLT will be from the first day of treatment until 30 days after receiving the first dose of leflunomide + decitabine. After 12 cycles (study duration) responding patients can continue progression with the assigned doses.

Staging studies, including bone marrow biopsy and complete blood counts will be performed within 45 days prior to study enrollment and again within 30 days after completing Cycle 3, Cycle 6, and Cycle 12 and within 30 days of discontinuing study treatment. A repeat bone marrow biopsy will be performed at the end of the study (Cycle 12). Patients will be followed every 3 months for 2 years after completion of study.

Study assessments will also include monitoring of all toxicities and adverse events. The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, will be used for grading adverse events and all toxicities

ELIGIBILITY:
Inclusion Criteria:

* Patient has pathologically confirmed diagnosis of MDS
* Patient has currently measurable disease meeting the following criteria:

  * Bone marrow biopsy with more than 5% blasts, AND
  * Absolute neutrophil count (ANC) less than 1,000/mcL, and/or platelet count less than 100,000/mcL and/or hemoglobin levels less than 10g/dL
* Patient has received one prior treatment with a DNA methyltransferase inhibitor (DNMTi), also commonly called hypomethylating agent (HMA). Patients whose MDS has IDH1/IDH2 mutations should have received at least one available IDH1/IDH2 inhibitor
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Patient has the following required baseline laboratory data (eligibility can be based on local lab results):

  * Total serum bilirubin level less than or equal to 2 times ULN
  * Estimated glomerular filtration rate (eGFR) greater than or equal to 45 mL/min/1.73 m2
* Patients who have undergone alloHSCT are eligible if they are more than 28 days post stem cell infusion, have no evidence of GVHD > Grade 1, and are more than a week off all immunosuppressive therapy
* If a female of childbearing potential, the patient has a negative serum or urine pregnancy test result within 7 days prior to the first dose of treatment. Women of non-childbearing potential are those who are postmenopausal greater than one year or who have had a bilateral tubal ligation or hysterectomy
* If female of childbearing potential or a male patient, patient agrees to use an effective contraceptive method from the time of informed consent, during the course of the study, and for 3 months following the last dose of treatment
* Patient understands and voluntarily signs the written informed consent prior to any study-specific procedures. A copy of the signed informed consent form will be retained by the treating institution

Exclusion Criteria:

* Patients receiving any other investigational agents, or concurrent chemotherapy or immunotherapy
* Patients with progression to acute myeloid leukemia
* Patients with other malignancies requiring systemic chemotherapy, immunotherapy or targeted therapy in the last four weeks
* Patients with uncontrolled bacterial, viral or fungal infections (undergoing appropriate treatment and with progression of clinical symptoms)
* Patients with active or latent tuberculosis
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that per Principal Investigator's judgment would limit compliance with study requirements
* Females who are pregnant or breast feeding
* Any other clinical conditions that in the opinion of the investigator would make the subject unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of incidences of regimen limiting toxicities (RLTs) | Date of first treatment up to 13 months
  Percentages of incidences of RLTs defined as:
  * A need to reduce the dose of one or both of the treatments
  * Discontinue the treatment due to dose limiting toxicities, AE/SAE
  * Be withheld at the discretion of the treating physician and on the basis of the expected adverse event

SECONDARY OUTCOMES:
Percentage of Complete Remission (CR) Rate (3rd cycle) | Within 30 days following the end of the 3rd cycle (cycle = 28 days)
  Percentage of patients achieving complete remission (CR) rate defined as bone marrow (BM): <5% myeloblasts (dysplasia may persist), and peripheral blood (PB): hemoglobin (Hb) ≥10 g/dL, platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L; blasts 0%. Full cytogenetic clearance of baseline abnormalities (complete cytogenetic response)
Percentage of Complete Remission (CR) Rate (6th cycle) | Within 30 days following the end of the 6th cycle (cycle = 28 days)
  Percentage of patients achieving complete remission (CR) rate defined as bone marrow (BM): <5% myeloblasts (dysplasia may persist), and peripheral blood (PB): hemoglobin (Hb) ≥10 g/dL, platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L; blasts 0%. Full cytogenetic clearance of baseline abnormalities (complete cytogenetic response)
Percentage of Complete Remission (CR) Rate (12th cycle) | Within 30 days of the end of the 12th cycle (cycle = 28 days)
  Percentage of patients achieving complete remission (CR) rate defined as bone marrow (BM): <5% myeloblasts (dysplasia may persist), and peripheral blood (PB): hemoglobin (Hb) ≥10 g/dL, platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L; blasts 0%. Full cytogenetic clearance of baseline abnormalities (complete cytogenetic response)
CR + complete remission with partial hematologic recovery (CRh) (3rd cycle) | Within 30 days following the end of the 3rd cycle (cycle = 28 days)
  Percentage of participants that achieve CR + complete remission with partial hematologic recovery (CRh) - defined as BM: <5% myeloblasts (dysplasia may persist) and PB: Not meeting criteria for CR or CRL, no Hb threshold required, platelets ≥50 × 109/L; neutrophils ≥0.5 × 109/L; blasts 0%
CR + complete remission with partial hematologic recovery (CRh) (6th cycle) | Within 30 days following the end of the 6th cycle (cycle = 28 days)
  Percentage of participants that achieve CR + complete remission with partial hematologic recovery (CRh) - defined as BM: <5% myeloblasts (dysplasia may persist) and PB: Not meeting criteria for CR or CRL, no Hb threshold required, platelets ≥50 × 109/L; neutrophils ≥0.5 × 109/L; blasts 0%
CR + complete remission with partial hematologic recovery (CRh) (12th cycle) | Within 30 days following the end of the 12th cycle (cycle = 28 days)
  Percentage of participants that achieve CR + complete remission with partial hematologic recovery (CRh) - defined as BM: <5% myeloblasts (dysplasia may persist) and PB: Not meeting criteria for CR or CRL, no Hb threshold required, platelets ≥50 × 109/L; neutrophils ≥0.5 × 109/L; blasts 0%
CR + CRh + complete remission with limited count recovery (CRL) including CR bilineage (CRbi) and CR unilineage (CRuni) (3rd cycle) | Within 30 days following the end of the 3rd cycle (cycle = 28 days)
  Percentage of participants that achieve CR + CRh + complete remission with limited count recovery (CRL) including CR bilineage (CRbi) and CR unilineage (CRuni) - defined as BM: <5% myeloblasts (dysplasia may persist), and PB: blasts 0%; CRuni: PB, not meeting CR but only 1 of the following: Hb ≥10 g/dL; platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L; CRbi: PB, not meeting CR but only 2 of the following: Hb ≥10 g/dL; platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L
CR + CRh + complete remission with limited count recovery (CRL) including CR bilineage (CRbi) and CR unilineage (CRuni) (6th cycle) | Within 30 days following the end of the 6th cycle (cycle = 28 days)
  Percentage of participants that achieve CR + CRh + complete remission with limited count recovery (CRL) including CR bilineage (CRbi) and CR unilineage (CRuni) - defined as BM: <5% myeloblasts (dysplasia may persist), and PB: blasts 0%; CRuni: PB, not meeting CR but only 1 of the following: Hb ≥10 g/dL; platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L; CRbi: PB, not meeting CR but only 2 of the following: Hb ≥10 g/dL; platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L
CR + CRh + complete remission with limited count recovery (CRL) including CR bilineage (CRbi) and CR unilineage (CRuni) (12th cycle) | Within 30 days following the end of the 12th cycle (cycle = 28 days)
  Percentage of participants that achieve CR + CRh + complete remission with limited count recovery (CRL) including CR bilineage (CRbi) and CR unilineage (CRuni) - defined as BM: <5% myeloblasts (dysplasia may persist), and PB: blasts 0%; CRuni: PB, not meeting CR but only 1 of the following: Hb ≥10 g/dL; platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L; CRbi: PB, not meeting CR but only 2 of the following: Hb ≥10 g/dL; platelets ≥100 × 109/L; neutrophils ≥1.0 × 109/L
Allogeneic hematopoietic stem cell transplant (alloHSCT) | Enrollment up to 3 years
  The percentage of participants that proceed to allogeneic hematopoietic stem cell transplant (alloHSCT).
Overall Survival (OS) | From first treatment up to 3 years
  Overall Survival (OS) defined for all patients of the trial; measured from the first day of receiving study drugs on the clinical trial to the date of death by any cause
Event-free survival (EFS) | From first treatment up to 3 years
  Event-free survival (EFS) defined for all patients of the trial; measured from the first day of receiving study drugs to the date of treatment failure, or relapse from CR or CRh or CRL, or death by any cause. Treatment is defined as failure to achieve CR or CRh or CRL after at least three cycles of treatment; the date of treatment failure is defined as date of marrow evaluation after the last course of treatment.
Relapse-free survival (RFS) defined only for patients achieving CR or CRh or CRL; | From the date of achievement of a CR/CRh/CRL up to 3 years
  Relapse-free survival (RFS) defined only for patients achieving CR or CRh or CRL; measured from the date of achievement of a CR/CRh/CRL until the date of relapse or death from any cause; RFS and disease-free survival (DFS) have been used with the same definition.
Progression to acute myeloid leukemia (AML) | Enrollment up to 3 years
  Percentage of participant progression to acute myeloid leukemia (AML)
Percentage of Red Blood Cell transfusion independence | Date of first treatment up to 3 years
  The percentage of participants that achieve the conversion from red blood cell transfusion dependence to transfusion independence. Transfusion Independence is defined as a period of time, usually 8 weeks, with no transfusion between first dose of study drug and the last dose of study drug + 30 days.

OTHER OUTCOMES:
Percentage Clonal Evolution | Enrollment up to 3 years
  Percentage of participants with clonal evolution. Defined as mutations in founding clone, expansion of subclone(s), and convergent clonal evolution of signaling gene mutations; assessed by chromosomal analysis, fluorescence in situ hybridization (FISH) and mutational analysis by next generation sequencing in bone marrow evaluation.
Percentage of platelet transfusion independence | Date of first treatment up to 3 years
  The percentage of participants that achieve the conversion from platelet transfusion dependence to transfusion independence (persons who transition from needing regular platelet transfusions to no longer requiring them).

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Sdrimas, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Cancer Institute, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chilakala S, Feng Y, Li L, Mahfouz R, Quteba E, Saunthararajah Y, Xu Y. Tracking Decitabine Incorporation into Malignant Myeloid Cell DNA in vitro and in vivo by LC-MS/MS with Enzymatic Digestion. Sci Rep. 2019 Mar 14;9(1):4558. doi: 10.1038/s41598-019-41070-y. PMID 30872721
- [Background] Qin F, Wu J, Chen F, Wei Y, Zhao Y, Jiang Z, Bai J, Yu H. Optimal, minimax and admissible two-stage design for phase II oncology clinical trials. BMC Med Res Methodol. 2020 May 20;20(1):126. doi: 10.1186/s12874-020-01017-8. PMID 32434577
- [Background] Zeidan AM, Platzbecker U, Bewersdorf JP, Stahl M, Ades L, Borate U, Bowen D, Buckstein R, Brunner A, Carraway HE, Daver N, Diez-Campelo M, de Witte T, DeZern AE, Efficace F, Garcia-Manero G, Garcia JS, Germing U, Giagounidis A, Griffiths EA, Hasserjian RP, Hellstrom-Lindberg E, Iastrebner M, Komrokji R, Kulasekararaj AG, Malcovati L, Miyazaki Y, Odenike O, Santini V, Sanz G, Scheinberg P, Stauder R, van de Loosdrecht AA, Wei AH, Sekeres MA, Fenaux P. Consensus proposal for revised International Working Group 2023 response criteria for higher-risk myelodysplastic syndromes. Blood. 2023 Apr 27;141(17):2047-2061. doi: 10.1182/blood.2022018604. PMID 36724453
- [Background] Kayamori K, Nagai Y, Zhong C, Kaito S, Shinoda D, Koide S, Kuribayashi W, Oshima M, Nakajima-Takagi Y, Yamashita M, Mimura N, Becker HJ, Izawa K, Yamazaki S, Iwano S, Miyawaki A, Ito R, Tohyama K, Lennox W, Sheedy J, Weetall M, Sakaida E, Yokote K, Iwama A. DHODH inhibition synergizes with DNA-demethylating agents in the treatment of myelodysplastic syndromes. Blood Adv. 2021 Jan 26;5(2):438-450. doi: 10.1182/bloodadvances.2020001461. PMID 33496740
- [Background] Santini V. How I treat MDS after hypomethylating agent failure. Blood. 2019 Feb 7;133(6):521-529. doi: 10.1182/blood-2018-03-785915. Epub 2018 Dec 13. PMID 30545832
- [Background] Stomper J, Rotondo JC, Greve G, Lubbert M. Hypomethylating agents (HMA) for the treatment of acute myeloid leukemia and myelodysplastic syndromes: mechanisms of resistance and novel HMA-based therapies. Leukemia. 2021 Jul;35(7):1873-1889. doi: 10.1038/s41375-021-01218-0. Epub 2021 May 6. PMID 33958699
- [Background] Jabbour E, Garcia-Manero G, Batty N, Shan J, O'Brien S, Cortes J, Ravandi F, Issa JP, Kantarjian H. Outcome of patients with myelodysplastic syndrome after failure of decitabine therapy. Cancer. 2010 Aug 15;116(16):3830-4. doi: 10.1002/cncr.25247. PMID 20564137
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Prebet T, Gore SD, Esterni B, Gardin C, Itzykson R, Thepot S, Dreyfus F, Rauzy OB, Recher C, Ades L, Quesnel B, Beach CL, Fenaux P, Vey N. Outcome of high-risk myelodysplastic syndrome after azacitidine treatment failure. J Clin Oncol. 2011 Aug 20;29(24):3322-7. doi: 10.1200/JCO.2011.35.8135. Epub 2011 Jul 25. PMID 21788559
- [Background] Zeidan AM, Stahl M, Hu X, Wang R, Huntington SF, Podoltsev NA, Gore SD, Ma X, Davidoff AJ. Long-term survival of older patients with MDS treated with HMA therapy without subsequent stem cell transplantation. Blood. 2018 Feb 15;131(7):818-821. doi: 10.1182/blood-2017-10-811729. Epub 2017 Dec 19. No abstract available. PMID 29259002
- [Background] Bartenstein M, Deeg HJ. Hematopoietic stem cell transplantation for MDS. Hematol Oncol Clin North Am. 2010 Apr;24(2):407-22. doi: 10.1016/j.hoc.2010.02.003. PMID 20359634
- [Background] Sekeres MA, Schoonen WM, Kantarjian H, List A, Fryzek J, Paquette R, Maciejewski JP. Characteristics of US patients with myelodysplastic syndromes: results of six cross-sectional physician surveys. J Natl Cancer Inst. 2008 Nov 5;100(21):1542-51. doi: 10.1093/jnci/djn349. Epub 2008 Oct 28. PMID 18957672